CLINICAL TRIAL: NCT01937455
Title: Safety and Immunogenicity Study of rAAV1-PG9DP Recombinant AAV Vector Coding for PG9 Antibody in Healthy Male Adults.
Brief Title: A Phase 1, Randomized, Blinded, Dose-escalation Study of rAAV1-PG9DP Recombinant AAV Vector Coding for PG9 Antibody in Healthy Male Adults.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IAVI A003/CHOP HVDDT 001; 2013-002268-14 (EudraCT Number); HHSN272201000021C (Other Grant/Funding Number: NIH contract)
Record Dates: First submitted 2013-09-04; First posted 2013-09-09 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; HIV vaccine; HIV prevention; AAV; PG9
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A (Experimental): rAAV1-PG9DP or placebo (v:p = 3:1)
  Interventions: Biological: rAAV1-PG9DP
- Group B (Experimental): rAAV1-PG9DP or placebo (v:p = 3:1)
  Interventions: Biological: rAAV1-PG9DP
- Group C/C1 (Experimental): rAAV1-PG9DP or placebo (v:p = 3:1 in Group C, and v:p = 9:3 in Group C1)
  Interventions: Biological: rAAV1-PG9DP
- Group D/D1 (Experimental): rAAV1-PG9DP or placebo (v:p = 3:1 in Group D, v:p = 4:1 in Group D1)
  Interventions: Biological: rAAV1-PG9DP

INTERVENTIONS:
Biological: rAAV1-PG9DP — 4x10^12 vg administered intramuscularly
  Arms: Group A
Biological: rAAV1-PG9DP — 4x10^13 vg administered intramuscularly
  Arms: Group B
Biological: rAAV1-PG9DP — 8x10^13 vg administered intramuscularly
  Arms: Group C/C1
Biological: rAAV1-PG9DP — 1.2x10^14 vg administered intramuscularly
  Arms: Group D/D1

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and immunogenicity of rAAV1-PG9DP when administered intramuscularly at different dose levels in healthy male adults.

DETAILED DESCRIPTION:
This study is a phase 1, randomized, blinded, dose-escalation study to evaluate the safety and tolerability of rAAV1-PG9DP when administered intramuscularly at 4x10^12 vg, 4x10^13 vg, 8x10^13 vg and 1.2x10^14 vg in healthy male adults.

Volunteers will be screened up to 42 days before injection and will be followed for 12 months after the single administration. It is anticipated that it will take approximately 13 months to enroll the study.

Volunteers will be randomly assigned investigational product (IP) or placebo within each of the dose groups described in the study design table above depending on which group is enrolling. Study staff and volunteers will be blinded only with respect to the allocation of placebo or IP. Blinding will not apply to the assignment of dosage levels.

Volunteers will be offered enrollment into a follow-up study at the research center when they have finished participating in the trial

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male.
2. 18 to 45 years of age.
3. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study.
4. In the opinion of the Principal Investigator or designee and based on Assessment of Informed Consent Understanding results, has understood the information provided and has provided informed consent.
5. Willing to undergo HIV testing, risk reduction counseling and receive HIV test results.
6. All sexually active males must be willing to use male condoms with all sexual partners (female or male) from the day of first injection until 3 months after the injection.
7. Willing to forgo donations of blood or any other tissues during the study and, for those who test HIV-positive due to vaccine-induced antibodies, until the anti-HIV antibody titers become undetectable.

Exclusion Criteria:

1. Confirmed HIV-1 or HIV-2 infection.
2. Any clinically relevant abnormality on history or examination including history of immunodeficiency or autoimmune disease; use of systemic corticosteroids, immunosuppressive, anticancer, or other medications considered significant by the investigator within the previous 6 months.
3. Any clinically significant acute or chronic medical condition that is considered progressive or in the opinion of the investigator makes the volunteer unsuitable for participation in the study.
4. Any of the following specific risk behaviour for HIV infection within 6 months prior to injection:

   * Unprotected sexual intercourse with a known HIV infected person or a partner known to be at high risk for HIV infection or a casual partner (i.e., no continuing established relationship)
   * Unprotected anal intercourse with another man (either insertive or receptive)
   * Three or more sexual partners
   * Engaged in sex work
   * Frequent excessive daily alcohol use or frequent binge drinking or chronic marijuana abuse or any other use of illicit drugs
   * History of newly-acquired syphilis, gonorrhea, non-gonococcal urethritis, HSV-2, chlamydia, epididymitis, proctitis, lymphogranuloma venereum, chancroid, or hepatitis B
5. Bleeding disorder that was diagnosed by a physician (e.g., factor deficiency, coagulopathy or platelet disorder that requires special precautions).
6. Clinically significant laboratory abnormalities.
7. Anti-AAV1 antibody level above the cut-off.
8. Receipt of live attenuated vaccine within the previous 60 days or planned receipt within 60 days after injection with IP; or receipt of other vaccine within the previous 14 days or planned receipt within 14 days after injection with IP (exception is live attenuated influenza vaccine within 14 days).
9. Receipt of blood transfusion or blood-derived products within the previous 3 months.
10. Participation in another clinical trial of an IMP currently, within the previous 3 months or expected participation during this study.
11. Prior receipt of another AAV vector, investigational HIV vaccine candidate, monoclonal antibody or polyclonal immunoglobulin (note: receipt of placebo in a previous HIV vaccine or monoclonal antibody trial will not exclude a volunteer from participation).
12. History of severe local or systemic reactogenicity to vaccines or infusions (e.g., anaphylaxis, respiratory difficulties, angioedema)
13. Psychiatric condition that compromises safety of the volunteer and precludes compliance with the protocol.
14. In the opinion of the Principal Investigator, it is not in the best interest of the volunteer to participate in the trial.
15. Seizure disorder: a participant who has had a seizure in the last 3 years.
16. ECG with clinically significant findings or features.
17. History of, or known active cardiovascular disease.
18. Have 3 or more of the following risk factors:

    * Hypertension diagnosed by a doctor
    * Hypercholesterolemia diagnosed by a doctor
    * Diabetes mellitus
    * Hyperglycemia diagnosed by a doctor
    * First degree relative (i.e., mother, father, brother, sister) who had a heart condition before the age of 50
    * Currently smoke cigarettes

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-09; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 12 months
  1. Proportion of volunteers with moderate or greater reactogenicity (i.e., solicited adverse events) during a 7 day follow-up period after the injection
  2. Proportion of volunteers with moderate or greater adverse events (i.e. unsolicited adverse events) including safety laboratory (biochemical, haematological) parameters, from the day of the injection up to 180 days post injection
  3. Proportion of volunteers with serious adverse events (SAEs) related to the IMP throughout the study period
  4. The proportion of volunteers in each group with Adverse Event of Special Interest, defined as adverse events potentially caused by antigen-antibody complexes or immune responses directed to cells producing the transgene

SECONDARY OUTCOMES:
Pharmacokinetics and Immunogenicity | 12 months
  To assess (qualitative and quantitative) immune responses elicited by the different dose levels.

CONTACTS AND LOCATIONS:
Overall Officials: David JM Lewis, Principal Investigator — Clinical Research Centre, Institute of Biosciences and Medicine, FHMS, University of Surrey
Locations (2):
- United Kingdom (2):
  - Surrey Clinical Research Centre, Guildford
  - Southampton Centre for Biomedical Research, Southampton

REFERENCES:
- [Derived] Libera M, Caputo V, Laterza G, Moudoud L, Soggiu A, Bonizzi L, Diotti RA. The Question of HIV Vaccine: Why Is a Solution Not Yet Available? J Immunol Res. 2024 Apr 8;2024:2147912. doi: 10.1155/2024/2147912. eCollection 2024. PMID 38628675
- [Derived] Priddy FH, Lewis DJM, Gelderblom HC, Hassanin H, Streatfield C, LaBranche C, Hare J, Cox JH, Dally L, Bendel D, Montefiori D, Sayeed E, Ackland J, Gilmour J, Schnepp BC, Wright JF, Johnson P. Adeno-associated virus vectored immunoprophylaxis to prevent HIV in healthy adults: a phase 1 randomised controlled trial. Lancet HIV. 2019 Apr;6(4):e230-e239. doi: 10.1016/S2352-3018(19)30003-7. Epub 2019 Mar 15. PMID 30885692
- See also: International AIDS Vaccine Initiative — http://www.iavi.org